CLINICAL TRIAL: NCT03299192
Title: Tai Chi for Chronic Low Back Pain in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34AT009052 (NIH)
Record Dates: First submitted 2017-05-31; First posted 2017-10-03 (Actual); Results first posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Back Pain Lower Back Chronic
MeSH Terms: interventions — Tai Ji

STUDY DESIGN:
Intervention Model Description: Comparison of Tai Chi to Health Education and to Usual Medical Care
Who Masked: Outcomes Assessor
Masking Description: Research Specialists will be unaware of study group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tai Chi (Experimental): twice weekly classes for 12 weeks and then weekly for 6 weeks, every other week for 6 weeks and monthly for 3 months
  Interventions: Behavioral: Tai Chi; Other: Usual Medical Care
- Health Education (Active Comparator): twice weekly classes for 12 weeks
  Interventions: Behavioral: Health Education; Other: Usual Medical Care
- Usual Medical Care (Active Comparator): the usual care to which participants are entitled by their health insurance
  Interventions: Other: Usual Medical Care

INTERVENTIONS:
Behavioral: Tai Chi — Yang Style Tai Chi
  Arms: Tai Chi
Behavioral: Health Education — Comprehensive Health Education relevant for Healthy Aging in Patients with Chronic Back Pain
  Arms: Health Education
Other: Usual Medical Care — Medications, PT, Complementary and Integrative Health and other miscellaneous treatments as appropriate.

SUMMARY:
There is a major gap in knowledge about safe and effective treatment options for older adults with chronic low back pain. This project will determine the feasibility of conducting a full-scale trial evaluating Tai Chi, a promising "mind-body" intervention that seems particularly well-suited for older adults with chronic low back pain.

DETAILED DESCRIPTION:
The ultimate goal of this project is to help fill the substantial gap in knowledge about safe and effective treatments for older adults with chronic low back pain. This deficiency is a particular problem because treatments that have been found safe and effective for younger adults may not be appropriate for an older population that is at higher risk of adverse effects and that may have different needs and treatment preferences. Tai Chi, which has been found effective for chronic back pain in younger adults, seems particularly well-suited for older adults with chronic low back pain because it includes multiple therapeutic elements, is gentle and has been found beneficial for a variety of health conditions more common to older adults. The goal of this project is to prepare the foundation for successfully conducting a full-scale trial evaluating the effectiveness of two doses of Tai Chi (Standard and Enhanced, which includes Standard + Maintenance Tai Chi) for improving chronic low back pain in older adults over the course of a year.

In the first phase of this study (Aim 1), the the Investigators will focus on finalization of a Standard Tai Chi protocol, development of the maintenance Tai Chi protocol and development of a credible attention control group. In the course of finalizing the feasibility trial documents, members of the research study team will work with patient partners (older adults with chronic low back pain) to adapt strategies for recruitment, adherence to Tai Chi, safety, and optimizing follow-up rates for this population and the Investigators will finalize the inclusion/exclusion criteria to maximize safety and generalizability.

After finalizing the key study components, the Investigators will conduct a randomized feasibility trial comparing Enhanced Tai Chi with Health Education and Usual Medical Care. Sixty-four older adults with cLBP - 65+ years of age will be randomized to the Enhanced (standard + maintenance) Tai Chi, to Health Education or to Usual Medical Care. Outcomes will be collected at 12, 26, and 52 weeks. The Investigators will evaluate the adequacy of key elements of the study developed in Aim 1 for inclusion in a full-scale trial. Finally, the research study team will conduct debriefing discussion groups with 30 trial participants to elicit their ideas for improving the procedures and protocols. This evaluation will address the overall feasibility of conducting a large trial and the value of including the Enhanced dose Tai Chi treatment arm.

If successful, this feasibility study will pave the way for conducting an adequately-powered randomized\ controlled trial evaluating the ability of Tai Chi to reduce the impact of chronic low back pain on older adults. In view of the absence of knowledge about clearly safe and effective treatments for this population, this line of research has the potential for substantially reducing the suffering of many Americans with back pain.

ELIGIBILITY:
Inclusion Criteria:

* • Be men or women at least 65 years of age

  * Have low back pain that has persisted for at least three months
  * Have had back pain on at least half the days in the last 6 months
  * Have at least moderate intensity low back pain
  * Have some activity limitations due to back pain
  * Be members of Kaiser Permanente Washington integrative health care system or have a regular source of health care and health insurance
  * Have normal cognition or only mild cognitive impairment
  * Be capable of understanding the study procedures and complying with them for the entire study period.
  * Live close enough to the class site for attendance to be practical
  * Give informed consent

Exclusion Criteria:

* • Have certain specific conditions of LBP

  * Prior lumbar spine surgery
  * Have sciatica, or scheduled visits to a neurosurgeon or orthopedic surgeon.
  * Receiving or seeking compensation for back pain
  * Red flags of serious underlying illness
  * Have practiced Tai Chi or yoga recently. Have other disabling conditions that might confound treatment effects
  * Conditions making consent or treatment difficult
  * Conditions making treatment unsafe or inappropriate
  * Unwillingness to give informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Washington Health Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tai Chi | Health Education | Usual Medical Care
Started | 28 | 12 | 17
Completed | 27 | 10 | 16
Not Completed | 1 | 2 | 1
Not completed — Fell before classes started | 1 | 0 | 0
Not completed — Other | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tai Chi | Health Education | Usual Medical Care | Total
Number analyzed (Participants) | 28 | 12 | 17 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 28 | 12 | 17 | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.2 (5.9) | 73.6 (5.5) | 71.8 (3.8) | 72.9 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 8 | 11 | 35
  Male | 12 | 4 | 6 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 1 | 8
  White | 21 | 9 | 11 | 41
  More than one race | 0 | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 12 | 17 | 57
Roland-Morris Disability Measure Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The score of the Roland-Morris Disability Questionnaire (RDMQ) is the total number of items checked, from a minimum of 0 to a maximum of 24, with a higher score indicating a higher experience of disability from back pain. The timeframe of the RMDQ is how a person feels within the last 7 days.
  units on a scale | 11.4 (4.3) | 11.7 (3.7) | 9.4 (4.2) | 10.8 (4.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Roland Morris Disability Questionnaire Score
Description: The score of the Roland-Morris Disability Questionnaire (RDMQ) is the total number of items checked, from a minimum of 0 to a maximum of 24, with a higher score indicating a higher experience of disability from back pain. The timeframe of the RMDQ is how a person feels within the last 7 days.
  Change was calculated as the value of the time point (3, 6, or 12 months) minus baseline
Time Frame: Baseline, 3, 6, 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tai Chi | Health Education | Usual Medical Care
Number analyzed (Participants) | 27 | 10 | 16
units on a scale
  3 Months | -4.38 [-5.81 to -2.96] | -0.12 [-2.58 to 2.93] | 0.18 [-2.58 to 2.93]
  6 Months | -3.64 [-5.64 to -1.65] | -1.92 [-3.73 to -0.11] | -2.39 [-4.79 to 0.01]
  12 Months | -5.20 [-7.11 to -3.29] | -0.82 [-3.04 to 1.40] | -2.89 [-4.74 to -1.04]
Statistical Analysis 1: Comparison: Tai Chi vs Health Education vs Usual Medical Care; Test type: Superiority; p = .001, GEE with Ancova features — This feasibility study is small and not designed to look at outcome statistics

ADVERSE EVENTS:
Time Frame: Adverse event information was collected over a 1-year period post-enrollment.
Arm/Group | Tai Chi | Health Education | Usual Medical Care
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/12 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/12 | 0/17
Other Adverse Events (participants affected / at risk) | 0/28 | 0/12 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT03299192/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT03299192/SAP_001.pdf
  • Informed Consent Form (2017-07-18): https://cdn.clinicaltrials.gov/large-docs/92/NCT03299192/ICF_002.pdf